CLINICAL TRIAL: NCT06609837
Title: 30-Second Sit-to-Stand Test as an Alternative Tool for Assessing Functional Capacity in Patients With Juvenile Idiopathic Arthritis
Brief Title: 30-Second Sit-to-Stand Test for Assessing Functional Capacity in Juvenile Idiopathic Arthritis
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nilay Arman, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: NArmann
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2024-09

CONDITIONS: Juvenile Idiopahtic Arthritis
Keywords: adolescents; Juvenile Idiopahtic Arthritis; functional capacity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Usability and Validity Group: In order to evaluate the usability of the 30SST, the validity of the test will be examined. In order to determine its validity in assessing functional capacity, the correlation of 6 MWT and 10SCT will be examined.
- Healthy Control Group: For analysis the difference between JIA and healthy control regarding the 30SST, 6MWT and 10SCT statistical analysis will be performed.

SUMMARY:
Juvenile Idiopathic Arthritis (JIA) is a heterogeneous, idiopathic, chronic inflammatory, rheumatic disease that is most common in childhood and is thought to involve immunological mechanisms in its etiopathogenesis. The physiology of children and adolescents is constantly changing due to the development and maturation of their systems. At the same time, the changes that this population shows, especially during the growth spurt and adolescence, can affect their performance in frequently used functional tests such as the 6-Minute Walk Test (6MWT). At the same time, it is emphasized that alternative tests are needed because the evaluation procedures of the 6MWT are not practical enough. The aim of this study is to investigate whether 30 Second Sit to Stand Test (30SST) is an alternative tool for assessing functional capacity in patients with JIA.

H0: 30SST is not an alternative tool for assessing functional capacity in patients with JIA.

H1: 30SST is an alternative tool for assessing functional capacity in patients with JIA.

The study will include 81 adolescent patients with oligoarticular/polyarticular JIA and 116 healthy adolescent between the ages of 12-18. The 6MWT, 30SST and 10 Stair Climb Test (10SCT) will be applied to the cases that meet the inclusion criteria to evaluate their functional capacity. Demographic data and test results of the participants will be recorded and evaluated with statistical analysis methods. We believe that alternative tests that can be used to evaluate functional capacity in patients with JIA will contribute to the literature as a result of this study.

ELIGIBILITY:
Inclusion Criteria:

* Being 12-18 years old for both groups
* Having been diagnosed with JIA at least 6 months ago at the Istanbul Medical Faculty Pediatric Rheumatology Clinic for Usability and Validity Group
* Having a diagnosis of Oligoarticular/Polyarticular JIA for Usability and Validity Group
* Volunteer to participate in the study for both groups

Exclusion Criteria:

* History of trauma or surgery affecting the musculoskeletal system within the last 6 months
* Having an additional chronic disease affecting the musculoskeletal system for both groups
* Having vision or hearing problems for both groups
* Having cognitive impairment at a level where the person cannot understand the commands given for both groups
* Having vision or hearing problems for both groups
* Having had a corticosteroid injection into the knee or ankle within the last week for both groups
* Difference in length in the lower extremities for both groups

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Individuals with JIA who come to Istanbul University Medical Faculty, Pediatric Rheumatology Clinic and meet the inclusion criteria for Usability and Validity Group Healthy adolescent participants aged 12-18 years
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test (6 MWT) | Time Frame: Baseline
  The 6MWT is a well-tolerated, easy-to-apply and simple test that shows the submaximal level of functional capacity. This test measures the distance that participants can walk quickly on a hard and flat surface in 6 minutes. Participants are rested in a chair near the starting position for at least 10 minutes before the test begins. Participants are instructed on how to perform the test. At the end of the test, the distance that participants walk in 6 minutes will be recorded in meters. The 6MWT will be used to evaluate the functional capacity of adolescents.
30 Second Sit to Stand Test (30SST) | Time Frame: Baseline
  The participant will be asked to sit in a chair with the back straight; Arms will be crossed at the wrists and held towards the chest. The participant will be encouraged to complete as many sit-ups as possible in 30 seconds. The participant will be instructed to sit up completely after each sit-up. The score will be noted as the total number of sit-ups in 30 seconds.
10 Stairs Climb Test (10SCT) | Time Frame: Baseline
  During the test, participants will be asked to climb 10 steps (14x28x120cm) as fast as possible. Step climbing times will be measured in seconds with a stopwatch. The 10SCT will be used to evaluate the functional capacity of adolescents.

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Arman, Assoc. Prof., Study Director — Istanbul University - Cerrahpasa; Asena Yekdaneh, MSc. Pt., Principal Investigator — Fenerbahçe University; Asya Albayrak, MSc. Pt., Principal Investigator — Istanbul University - Cerrahpasa; Fatma Gül Demirkan, Dr., Principal Investigator — Istanbul University; Özlem Akgün, Assoc. Prof., Principal Investigator — Istanbul University; Nuray Aktay Ayaz, Prof., Principal Investigator — Istanbul University
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No